CLINICAL TRIAL: NCT05922228
Title: Effects of Neural Flossing With and Without Proprioceptive Neuromuscular Facilitation on Pain, Range of Motion and Disability in Patients With Lumbar Radiculopathy.
Brief Title: Effects of Neural Flossing and PNF on Lumbar Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0212
Record Dates: First submitted 2023-06-06; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Lumbar Radiculopathy
Keywords: Disability; Lumbar; PNF; Neural flossing; pain
MeSH Terms: conditions — Radiculopathy; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural flossing with proprioceptive neuromuscular facilitation (Experimental): nerve flossing technique protocol along with contract relax technique of proprioceptive neuromuscular facilitation is used
  Interventions: Other: neural flossing with proprioceptive neuromuscular facilitation
- Neural flossing without proprioceptive neuromuscular facilitation (Active Comparator): only nerve flossing technique protocol is used
  Interventions: Other: Neural flossing without proprioceptive neuromuscular facilitation

INTERVENTIONS:
Other: neural flossing with proprioceptive neuromuscular facilitation — neural flossing technique for 5minutes, 10 repetitions×1 set, 3 days/week contract relax technique of proprioceptive neuromuscular facilitation for 5 minutes, 10 repetitions ×1 set, 3 days/week total of 15 sessions were given as 3 sessions/week up to 5 weeks, each session consisting of 10 minutes
  Arms: Neural flossing with proprioceptive neuromuscular facilitation
Other: Neural flossing without proprioceptive neuromuscular facilitation — neural flossing technique for 5minutes, 10 repetitions×1 set, 3 days/week total of 15 sessions were given as 3 sessions/week up to 5 weeks, each session consisting of 5 minutes
  Arms: Neural flossing without proprioceptive neuromuscular facilitation

SUMMARY:
the goal of this clinical trial is to determine the effects of neural flossing with and without proprioceptive neuromuscular facilitation on pain, range of motion and disability in patients with lumbar radiculopathy. the main question it aim to answer is :- Does proprioceptive neuromuscular facilitation added benefit when combined with neural flossing to pain, range of motion and disability in lumbar radiculopathy patients? Research will compare the neural flossing group with the group receiving neural flossing with proprioceptive neuromuscular facilitation to see if there is any difference in the outcomes.

DETAILED DESCRIPTION:
Lumbar radiculopathy is a mutual condition amongst persons presenting to a spinal physician for consultation. Lumbar radiculopathy is a term used to describe the pain that is started in low back and radiated along the nerve root. The patient mostly complains from a low back pain that radiates toward the legs. Symptoms may include radiating pain, weakness, hypo-reflexia and gait abnormalities. The pain is caused by the neurological manifestations of a compressive force along a specific nerve route. The main cause of radiculopathy is compression or irritation of nerve root exited from spinal cord. Lumbar radiculopathy can affect anyone regardless of their age, gender, race and geographical locality. About 40% people developed low back pain at some points in their life and out of them 3-5% population developed lumbar radiculopathy.

A study conducted to find out the influence of nerve flossing technique on acute sciatica and hip range of motion with sample size of 32. It was concluded that as a result of nerve flossing technique since no statistically significant changes occurred between the two groups. Hence, for effective reduction of sciatic pain and possible improvement in hip range of motion, nerve flossing technique should be combined with conventional physiotherapy. A study conducted on mobilization of Neurodynamic system using proprioceptive neuromuscular facilitation (PNF) decrease pain and increase mobility in lower extremities and spine suggested that PNF based rehabilitation approach results in improvement of pain, nerve mobility and balance.it also has positive effects by supplying oxygen to nerve, increase nerve mobility and decrease pain.

Some studies have been done testing the effects of neural flossing technique and PNF techniques individually as a treatment option for lumbar radiculopathy. But, up to the researcher's knowledge there is little literature on comparing both treatments with respect to pain, range of motion and disability in lumbar radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-50 years.
* Both males and females.
* Pain intensity is 4 out of 10 on numeric pain rating scale.
* History of radiculopathy for more than 3 weeks.
* Pain radiating below to knee.

Exclusion Criteria:

* Cognitive impairment.
* Using pain modulating medicines.
* Patients with comorbidities.
* Pain radiating above to knee.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 5 weeks
  It is a common pain screening tool use to assess the severity of pain at moment time. It is 0-10 scale where 0 means no pain and 10 means worst pain imaginable.
Goniometer | 5 weeks
  It is an instrument used to measure the available range of motion at joints. It is most commonly used tool to measure the range of motion of joints by physiotherapists.
Oswestry Disability Index (ODI) | 5 weeks
  The Oswestry Disability Index (ODI) is the most commonly used outcome-measure questionnaire for low back pain in a hospital setting. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability.

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, phd, Principal Investigator — Riphah International University
Locations (1):
- Aziz Bhatti Shaheed Teaching Hospital, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoenfeld AJ, Laughlin M, Bader JO, Bono CM. Characterization of the incidence and risk factors for the development of lumbar radiculopathy. J Spinal Disord Tech. 2012 May;25(3):163-7. doi: 10.1097/BSD.0b013e3182146e55. PMID 22543563
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Ghasabmahaleh SH, Rezasoltani Z, Dadarkhah A, Hamidipanah S, Mofrad RK, Najafi S. Spinal Manipulation for Subacute and Chronic Lumbar Radiculopathy: A Randomized Controlled Trial. Am J Med. 2021 Jan;134(1):135-141. doi: 10.1016/j.amjmed.2020.08.005. Epub 2020 Sep 13. PMID 32931763
- [Background] Senol D, Erdem C, Canbolat M, Toy S, Karatas T, Baykara RA, Ozbag D, Akyurek G. Comparison of the effects of conventional physiotherapy and proprioception exercises on pain and ankle proprioception in patients with lumbar radiculopathy. J Back Musculoskelet Rehabil. 2022;35(2):421-428. doi: 10.3233/BMR-200361. PMID 34308899
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Kahlaee AH, Ghamkhar L, Arab AM. The Association Between Neck Pain and Pulmonary Function: A Systematic Review. Am J Phys Med Rehabil. 2017 Mar;96(3):203-210. doi: 10.1097/PHM.0000000000000608. PMID 27610549
- [Background] Luoto S, Taimela S, Hurri H, Aalto H, Pyykko I, Alaranta H. Psychomotor speed and postural control in chronic low back pain patients A controlled follow-up study. Spine (Phila Pa 1976). 1996 Nov 15;21(22):2621-7. doi: 10.1097/00007632-199611150-00012. PMID 8961450
- [Background] Newcomer KL, Jacobson TD, Gabriel DA, Larson DR, Brey RH, An KN. Muscle activation patterns in subjects with and without low back pain. Arch Phys Med Rehabil. 2002 Jun;83(6):816-21. doi: 10.1053/apmr.2002.32826. PMID 12048661
- [Background] Barden JM, Balyk R, Raso VJ, Moreau M, Bagnall K. Dynamic upper limb proprioception in multidirectional shoulder instability. Clin Orthop Relat Res. 2004 Mar;(420):181-9. doi: 10.1097/00003086-200403000-00025. PMID 15057095
- [Background] Gunning E, Uszynski MK. Effectiveness of the Proprioceptive Neuromuscular Facilitation Method on Gait Parameters in Patients With Stroke: A Systematic Review. Arch Phys Med Rehabil. 2019 May;100(5):980-986. doi: 10.1016/j.apmr.2018.11.020. Epub 2018 Dec 22. PMID 30582917